CLINICAL TRIAL: NCT04858867
Title: Reinducing Radioiodine-sensitivity in Radioiodine-refractory Differentiated Thyroid Cancer Using Lenvatinib (RESET)
Brief Title: Reinducing Radioiodine-sensitivity in Radioiodine-refractory DTC Using Lenvatinib (RESET)
Acronym: RESET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, HW Kapiteijn, Medical Oncologist, Associate Professor Research and Treatment of Rare Cancers, Leiden University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P20.096
Record Dates: First submitted 2021-04-09; First posted 2021-04-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Study procedures
  * Lenvatinib during week 1-12
  * rhTSH-stimulated I-124 dosimetry at week 0, 6 and 12
  * rhTSH-stimulated I-131 therapy at week 13 (if eligible)
  * Intra-therapeutic I-131 dosimetry at week 13 (if eligible)
  * Biopsy at week 0 and 6
  * F-18 FDG PET/CT at week 0, 6, 12, 24 and 36
  * Tg levels at week 0, 6, 12, 24 and 36
  * QoL assessment at week 0, 6, 12, 24 and 36
  Interventions: Radiation: rhTSH-stimulated I-124 dosimetry; Radiation: Intra-therapeutic I-131 dosimetry
- Cohort 2 (Other): Study procedures (in case of 12-wk lenvatinib):
  * Lenvatinib during week 1-12
  * rhTSH-stimulated I-124 dosimetry at week 0 and 12
  * rhTSH-stimulated I-131 therapy at week 13 (if eligible)
  * Intra-therapeutic I-131 dosimetry at week 13 (if eligible)
  * Biopsy at week 0 and 6
  * F-18 FDG PET/CT at week 0, 12, 24 and 36
  * Tg levels at week 0, 6, 12, 24 and 36
  * QoL assessment at week 0, 6, 12, 24 and 36
  Study procedures (in case of 6-wk lenvatinib)
  * Lenvatinib during week 1-6
  * rhTSH-stimulated I-124 dosimetry at week 0 and 6
  * rhTSH-stimulated I-131 therapy at week 13 (if eligible)
  * Intra-therapeutic I-131 dosimetry at week 13 (if eligible)
  * Biopsy at week 0 and 6
  * F-18 FDG PET/CT at week 0, 6, 12, 24, 30 and 36
  * Tg levels at week 0, 6, 12, 24, 30 and 36
  * QoL assessment at week 0, 6, 12, 24, 30 and 36
  Interventions: Radiation: rhTSH-stimulated I-124 dosimetry; Radiation: Intra-therapeutic I-131 dosimetry

INTERVENTIONS:
Radiation: rhTSH-stimulated I-124 dosimetry — Preparation:
  * Low iodine diet 7 days prior to I-124 ingestion until 24 hours post-ingestion
  * Thyrogen injections 24 and 48h prior to I-124 ingestion
  Procedures following Jentzen et al:
  * Ingestion of capsule with 37±10% MBq I-124
  * I-124 PET/CT at 24 and 96h post-ingestion
  * Blood draws at 2, 24 and 96h post-ingestion
  * Whole body counting at 2, 24 and 96h post-ingestion
Radiation: Intra-therapeutic I-131 dosimetry — Procedures following EANM guidelines:
  * I-131 SPECT/CT at 2, 6, 24, 96 and 144h post-ingestion
  * Blood draws at 2, 6, 24, 96 and 144h post-ingestion
  * Whole body counting at 2, 6, 24, 96 and 144h post-ingestion

SUMMARY:
This is a single-centre open label phase II study evaluating the effect of lenvatinib treatment for restoring radioiodine uptake and retention in radioiodine-refractory (RAI-R) thyroid cancer to warrant I-131 therapy.

DETAILED DESCRIPTION:
RAI-R DTC patients starting standard-of-care lenvatinib treatment will be included in this study. Prior to lenvatinib treatment, patients will undergo I-124 PET/CT to quantify RAI uptake and retention at baseline. The first half of the intended sample size (cohort 1) will be treated with lenvatinib for a total of 12 weeks. After 6- and 12-week treatment, patients will undergo I-124 PET/CT dosimetry to evaluate the redifferentiation effect, assess expected absorbed lesion doses and maximum tolerable activity. Results between 6- and 12-week lenvatinib treatment will be compared to select the lenvatinib treatment duration that leads to highest extent of redifferentiation. The next patients (cohort 2) will then receive lenvatinib for either 6 or 12 weeks.

Patients will undergo subsequent I-131 therapy if a clinically meaningful lesion dose is expected and toxicity is deemed acceptable. For all patients eligible for I-131 therapy, lenvatinib is discontinued prior to administration of I-131 and intra-therapeutic I-131 SPECT dosimetry will be performed for dose verification. Patients who are not eligible for I-131 therapy, will continue lenvatinib treatment at the discretion of the treating physician.

Biopsies are performed at baseline and after 6-week lenvatinib treatment to evaluate alterations at the transcriptional and translational level in biopted tumor lesions. Patients will be followed up according to current guidelines for a total of 9 months after initiating lenvatinib treatment. Metabolic and biochemical response will be assessed using F-18 FDG PET/CT and Tg levels, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* Histologically or cytologically confirmed DTC (including papillary, follicular or Hürthle Cell carcinoma)
* Progressive (biochemical or anatomic) disease for which lenvatinib is started as standard treatment at the discretion of the treating physician
* Measurable disease at baseline imaging (F-18 FDG PET) according to the definition of the Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) 1.0 with at least one lesion ≥1.0 cm in the longest diameter for a non-lymph node or ≥1.5 cm in the short axis for a lymph node.
* RAI-R disease on structural imaging, defined as any one of the following:

  * Metastatic lesions that are not RAI-avid on a diagnostic or intra-therapeutic RAI scanperformed prior to enrolment in the current study
  * RAI-avid metastatic lesions which remained stable in size or progressed according to RECIST 1.1 criteria despite RAI treatment. Absence of response is observed during 6-9 months after high dose I-131 therapy.
* No recent treatment for thyroid cancer:

  * No prior I-131 therapy is allowed <6 months prior to initiation of therapy on this protocol (a diagnostic study using <400 MBq of I-131 is not considered 131I therapy)
  * No external beam radiation therapy is allowed <4 weeks prior to initiation of therapy on this protocol. (Previous treatment with radiation for any indication is allowed if the investigator judges that the previous radiation does not significantly compromise patient safety on this protocol)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (or Karnofsky ≥60%)
* Life expectancy ≥3 months
* Ability to swallow and retain orally-administered medication and no clinically significant gastrointestinal abnormalities that may alter absorption
* Creatinine ≤1.5 mg/dL (≤133 µmol/L) or estimated glomerular filtration rate (eGFR) (using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) ≥50 mL/min/1.73m2 or 24-hour urine creatinine clearance ≥50 mL/min/1.73m2
* Adequate blood coagulation function as evidenced by an international normalized ratio (INR) ≤1.5
* Adequate bone marrow function with:

  * Absolute neutrophil count ≥1.5*10^9 /L
  * Hemoglobin ≥9 g/dL (5.6 mmol/L)
  * Platelets ≥100*10^9 /L
* Adequate liver function with

  * Albumin ≥25 g/L
  * Total bilirubin <1.5x institutional upper limit of normal (ULN) with an exception for patients with Gilbert's syndrome
  * Aspartate aminotransferase and alanine aminotransferase ≤3x institutional ULN (≤5x ULN if subject has liver metastases)
* Negative pregnancy test within 7 days prior to starting the study for premenopausal women. Women can be included without pregnancy test if they are either surgically sterile or have been postmenopausal for ≥1 year.
* Sexually active women of childbearing potential must agree to use a highly effective method of contraception during the study and for at least 6 months after the last study treatment administration.Sexually active males patients must agree to use condom during the study and for at least 6 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception. Effective methods of contraception are defined as those, which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intrauterine devices). At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Concomitant or previous malignancies within the last 3 years. Patients are eligible for this study if they have been disease-free of the previous malignancy for at least 3 years, have a history of completely resected non-melanoma skin cancer and/or have indolent secondary malignancies.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* Evidence of cardiovascular risk including any of the following:

  * Clinically relevant arrhythmias
  * Acute coronary syndromes, severe/unstable angina
  * Symptomatic congestive heart failure
* Use of other investigational drugs within 28 days preceding the first dose of treatment in this study or during the study
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lenvatinib and/or to Thyrotropin alfa (human recombinant thyrotropin) or other known contents of the two drugs.
* Inability to follow a low iodine diet or requiring medication with high content in iodide (e.g. amiodarone)
* Patients who received iodinated intravenous contrast as part of a radiographic procedure within 6-8 weeks of study registration. Patients are eligible for this study if urinary iodine analysis reveals that the excess iodine has been adequately cleared after the last intravenous contrast administration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant, lactating or breast feeding women
* Any medical or other condition that in the opinion of the investigator(s) would preclude the participation in a clinical study
* Unwillingness or inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Fraction of RAI-R thyroid cancer patients who are eligible for I-131 therapy after 6- or 12-week lenvatinib treatment | 2-3 months after completed inclusion of all study participants
  Patients are deemed eligible for I-131 therapy if the therapeutic activity (max. 7.4 GBq) will lead to (1) an expected absorbed dose >20 Gy in at least one lesion, (2) a blood dose <2 Gy and (3) whole body retention <3.0 or 4.4 GBq at 48h post-ingestion in presence or absence of diffuse pulmonary metastases, respectively.

SECONDARY OUTCOMES:
Extent of RAI uptake at baseline and after 6- or 12-week lenvatinib | 0, 6, 12 weeks after inclusion
  Assessing expected absorbed dose [Gy] per lesion or critical organ using I-124 PET/CT, whole body counting and blood sampling
Optimal duration of lenvatinib treatment for maximum redifferentiation to occur | 3 months after completed inclusion of cohort 1
  Either 6 of 12 weeks after comparing (1) fraction of patients eligible for I-131 therapy, (2) expected absorbed dose [Gy] per lesion or critical organ and (3) toxicity incidence and severity
Extent of RAI uptake after I-131 therapy | 7 or 12 weeks after inclusion
  Assessing expected absorbed dose [Gy] per lesion or critical organ using intra-therapeutic I-131 SPECT/CT, whole body counting and blood sampling
Metabolic treatment response using F-18 FDG PET | 0, 6, 12, 24, 30, 36 weeks after inclusion
  Metabolic response will be assessed using PERCIST v1.0. Tumor response is defined as complete response, partial response, stable response or progressive disease.
Unstimulated (TSH suppressed) thyroglobulin levels | 0, 6, 12, 24, 30, 36 weeks after inclusion
  Assessment of biochemical treatment response
Overall survival at 36 weeks after initation of lenvatinib | 9 months after inclusion
Best objective response at 36 weeks after initation of lenvatinib | 9 months after inclusion
Progression free survival at 36 weeks after initation of lenvatinib | 9 months after inclusion
Incidence and severity of toxicities according to CTCAE 5.0 | during 0-9 months after inclusion
Quality of life using standardized questionnaire ThycaQoL | 0, 6, 12, 24, 30, 36 weeks after inclusion
Quality of life using standardized questionnaire RAND36 | 0, 6, 12, 24, 30, 36 weeks after inclusion
Quality of life using standardized questionnaire EQ5D5L | 0, 6, 12, 24, 30, 36 weeks after inclusion
Quality of life using standardized questionnaire Distress thermometer | 0, 6, 12, 24, 30, 36 weeks after inclusion

OTHER OUTCOMES:
NIS expression in biopted tumor lesion(s) at baseline and 6 weeks after lenvatinib | 0 and 6 weeks after inclusion
  An explorative endpoint of this study is to evaluate alterations at the transcriptional and translational level in biopted tumour lesions before and after lenvatinib treatment and to determine whether treatment response is related to genetical profiles

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kapiteijn, MD, PhD, Principal Investigator — LUMC; Dennis Vriens, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Dotinga M, Vriens D, van Velden F, Heijmen L, Nagarajah J, Hicks R, Kapiteijn E, de Geus-Oei LF. Managing radioiodine refractory thyroid cancer: the role of dosimetry and redifferentiation on subsequent I-131 therapy. Q J Nucl Med Mol Imaging. 2020 Sep;64(3):250-264. doi: 10.23736/S1824-4785.20.03264-1. PMID 32744039
- [Background] Dotinga M, Vriens D, van Velden FHP, Stam MK, Heemskerk JWT, Dibbets-Schneider P, Pool M, Rietbergen DDD, de Geus-Oei LF, Kapiteijn E. Reinducing Radioiodine-Sensitivity in Radioiodine-Refractory Thyroid Cancer Using Lenvatinib (RESET): Study Protocol for a Single-Center, Open Label Phase II Trial. Diagnostics (Basel). 2022 Dec 14;12(12):3154. doi: 10.3390/diagnostics12123154. PMID 36553163